CLINICAL TRIAL: NCT00028652
Title: Treament of Spontaneous Tumor Metastases With IL-12 DNA (NSC #709933): A Phase IB Trial
Brief Title: Interleukin-12 Gene Therapy in Treating Patients With Skin Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000069115; P30CA014520 (NIH); WCCC-CO-9771; WCCC-HSC-1998-257; NCI-T98-0025
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2015-09

CONDITIONS: Metastatic Cancer
Keywords: skin metastases
MeSH Terms: conditions — Neoplasm Metastasis

INTERVENTIONS:
Biological: interleukin-12 gene

SUMMARY:
RATIONALE: Inserting the gene for interleukin-12 into a person's skin tumor cells may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-12 gene therapy in treating patients who have skin metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of interleukin-12 gene in patients with spontaneous skin metastases.
* Determine the antitumor immune response in patients treated with this regimen.
* Compare the toxicity of this regimen administered for 1 week vs 2 weeks in these patients.
* Compare the local and systemic antitumor response in patients treated with this regimen administered for 1 week vs 2 weeks.

OUTLINE: Patients are stratified according to number of tumor sites (1 vs 2 vs 3 or more). Patients are assigned to 1 of 2 treatment arms.

* Group A: Patients receive interleukin-12 gene intratumorally over 5 minutes on days 1, 3, and 5.
* Group B: Patients receive IL-12 gene intratumorally over 5 minutes on days 1, 3, 5, 8, 10, and 12.

Patients with stable or responding disease may receive 1 subsequent course beginning on day 29.

Patients are followed at 3, 6, and 12 months.

PROJECTED ACCRUAL: A total of 12 patients (6 per treatment group) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid malignancy

  * Surgically or medically incurable disease
  * No standard chemotherapy or radiotherapy exists for this disease
* Tumor of at least 0.5 cm but no more than 2.5 cm infiltrating into or underlying the skin

  * Cutaneous metastases, subcutaneous metastases, or tumor-involved lymph nodes that are easily palpable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 80,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* HIV negative
* No active infections requiring antibiotic, antiviral, or antifungal treatment
* No other active malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 month since prior immunotherapy
* No concurrent colony-stimulating factors

Chemotherapy:

* See Disease Characteristics
* At least 1 month since prior chemotherapy

Endocrine therapy:

* At least 1 month since prior steroids (other than intermittent use as an antiemetic or topical agent)
* No concurrent steroids

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy to vaccine site allowed provided there is documentation of progressive disease

Surgery:

* See Disease Characteristics
* No prior organ allografts

Other:

* No other concurrent antineoplastic therapy
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: David M. Mahvi, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States